CLINICAL TRIAL: NCT02156141
Title: High Intensity Training in Patients With Spinal and Bulbar Muscular Atrophy
Acronym: HIT in Kennedy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karen Brorup Heje Pedersen (Other)
Responsible Party: Sponsor-Investigator, Karen Brorup Heje Pedersen, Bachelor in medicine, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H-4-2014-035
Record Dates: First submitted 2014-06-04; First posted 2014-06-05 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Spinal and Bulbar Muscular Atrophy; Healthy Subjects
Keywords: Kennedy's disease; Spinal and bulbar muscular atrophy; High Intensity Training; High Intensity Interval Training; HIT; HIIT; Training; Exercise; 10-20-30
MeSH Terms: conditions — Bulbo-Spinal Atrophy, X-Linked; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Supervised high intensity training (Experimental): 8 weeks of supervised high intensity training, 10 minutes, 3 times a week (once a week supervised) on a cycle ergometer followed by 8 weeks of unsupervised optional training.
  Participants: Patients with Kennedy's disease or healthy control subjects (individually matched with patients).
  Participants: Patients with Kennedys disease and healthy control subjects.
  Interventions: Other: Supervised high intensity training; Other: Optional training
- Unsupervised High intensity training (Experimental): 8 week control period with no training followed by 8 weeks of unsupervised high intensity training on a cycle ergometer.
  Participants: Patients with Kennedy's disease.
  Interventions: Other: Control period; Other: Unsupervised High intensity training

INTERVENTIONS:
Other: Supervised high intensity training — 8 weeks of supervised training
  Arms: Supervised high intensity training
Other: Optional training — 8 weeks of optional training on cycle ergometer. No program needs to be followed. Participant decides whether they want to keep training or not.
  Arms: Supervised high intensity training
Other: Control period — 8 weeks with no training.
  Arms: Unsupervised High intensity training
Other: Unsupervised High intensity training — 8 weeks of unsupervised high intensity training.
  Arms: Unsupervised High intensity training

SUMMARY:
We want investigate if high intensity training can increase daily functionality without causing muscle damage in patients Spinal and Bulbar Muscular Atrophy . We want to study if there is a difference in effect with supervised and unsupervised training. Furthermore we want to study if a supervised training program will motivate participants to continue training by the end of the program.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Spinal and bulbar muscular atrophy or
* Healthy control subjects matched individually with participating patients on age, sex, BMI and activity level.

Exclusion Criteria:

* More than 1 hour of fitness weekly before inclusion
* Other disease possibly confounding the results
* Pregnancy or breastfeeding
* Participations in other scientific studies wich could influence on the results during the last 30 days before inclusion.
* Physical and/or mental conditions preventing participating in the study protocol.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06-01 (Actual)

PRIMARY OUTCOMES:
Incremental test | Baseline, week 6, week 11, week 18
  Primary outcome is changes from baseline in maximal oxygen consumption and maximal workload after a 8 week supervised training program followed by a 8 week non-supervised optional training period.
  during and after 8 weeks of High Intensity Training on a cycle ergometer. The outcome is measured by an incremental test on a cycle ergometer.

SECONDARY OUTCOMES:
Functional test | Baseline, week 6, week 11, week 18.
  Changes from baseline to end of training in muscle strength measured by handhold dynamometry, in 6 minute walk-test and in 5 time sit-to-stand test is secondary outcome.
Self-rated muscle fatigue, muscle pain and activity level | Every day in week 1-11
  Self-rated muscle fatigue, muscle pain (VAS) and activity level is noted every day in diary in the two "run-in" weeks (baseline data) and thereafter every day in the 8 weeks training program. Changes from baseline is a secondary outcome.
Serum concentrations of Creatine Kinase (CK) | Baseline, Week 3,4,5,6,7,8,9,10,11, week 18.
  Serum concentrations of Creatine Kinase (CK) as a measurement of muscle damage. Blood samples are taken at every test day wich is the same for patient group 1 and healthy controls.
  In patient group 2 blood samples are taken at baseline, week 6, week 11 and week 18-
Activity level | Baseline, week 10 and week 18.
  Activity levels are measured by using a pedometer for a week at baseline, week 10 and week 18. Changes from baseline is a secondary outcome.

OTHER OUTCOMES:
Serum IGF-1 | Baseline, week 11, week 18.
  Changes in serum IGF-1 from baseline to week 11 and 18.

CONTACTS AND LOCATIONS:
Locations (1):
- Neuromuscular Research Unit, Copenhagen, Denmark

REFERENCES:
- See also: Website of Neuromuscular Research Unit, Rigshospitalet, Denmark. — http://www.neuromuscular.dk